CLINICAL TRIAL: NCT05311566
Title: Effectiveness and Safety of Camrelizumab Combined With Concurrent Chemoradiotherapy for FIGO IB2-IIIB Cervical Cancer: A Single-center, Single-arm, Open-phase II Clinical Study
Brief Title: PD-1 Antibody Plus Chemoradiotherapy for IB2-IIIB Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMURADIO3
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Cervical Carcinoma; Chemoradiotherapy; Anti-programmed Cell Death Receptor 1; Immunotherapy; Immune Checkpoint Inhibitor; Survival Outcomes; Adverse Events; Early Stage Cervical Cancer; Locally Advanced Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — camrelizumab; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with primary IB2-IIIB cervical cancer (Experimental): Patients with primary IB2-IIIB cervical cancer, including squamous carcinoma, adenocarcinoma, and adenosquamous carcinoma.
  Interventions: Combination Product: Camrelizumab plus Concurrent chemoradiotherapy

INTERVENTIONS:
Combination Product: Camrelizumab plus Concurrent chemoradiotherapy — Participants will be given intravenous administration of Camrelizumab (200mg，every 2 weeks),Cisplatin(40mg/m²，everyweek) and Radiotherapy. After completing 6~8weeks of concurrent chemoradiation, the Participants will continue to use camrelizumab as maintenance therapy until disease progression or unacceptable toxicity.

SUMMARY:
This study is a single-center, single-arm, open-phase II clinical study, the main purpose of which is to evaluate the effectiveness and safety of camrelizumab combined with concurrent chemoradiotherapy for early and locally advanced cervical cancer, i.e., FIGO 2018 IB2-IIIB cervical cancer. Eligible subjects will be given cisplatin and radiotherapy, for 6-8 weeks, camrelizumab repeated every 14 days until disease progression, toxicity intolerance, or other reasons specified in the protocol. Subjects who finished treatment entered the safety follow-up or survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed cervical adenocarcinoma, cervical squamous cell carcinoma, or cervical adenosquamous carcinoma and FIGO2018 IB2 to IIIB；
2. Have not received radiotherapy, chemoradiotherapy or other'system therapy for,cervical,cancer in the past.
3. With measurable tumor lesions (meet RECIST 1.1 standard).
4. Age≥18 years old when signing the informed consent, female.
5. ECOG PS: 0-2 points.
6. Expected survival time > 6 months.
7. According with lab testing criteria in the protocol.
8. Ability and willingness to comply with research and follow-up procedures.
9. Females of childbearing potential must agree to use adequate contraception throughout the study period and for 6 months after the end of treatment.
10. The patients voluntarily joined the clinical study and signed the informed consent, with good compliance and follow-up.

Exclusion Criteria:

1. Have previously received an anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, or anti-CTLA-4 antibody (or any other antibody that acts on T cell costimulation or checkpoint pathways);
2. Have a clear history of allergies, and may have potential allergies or intolerances to the study drug and its similar biological agents.
3. Participated in clinical trials of other antitumor drugs within 4 weeks before the first dose, or planned to receive live attenuated vaccines within 4 weeks before the first dose or during the study.
4. Other malignant tumors have occurred within 5 years (except for adequately treated cutaneous squamous cell carcinoma or controlled cutaneous basal cell carcinoma).
5. Use immunosuppressive medications, excluding nasal and inhaled corticosteroids or physiologic doses of systemic steroids (no more than 10 mg/day prednisolone or other corticosteroids at equivalent doses),within 14 days of first use of camrelizumab.
6. Symptomatic advanced patients with visceral dissemination who are at short-term risk of life-threatening complications (including uncontrolled massive exudates [thoracic, pericardium, abdominal], pulmonary lymphangitis and more than 30% patients with liver involvement).
7. Presence or history of any active autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma in childhood have been completely relieved, no need for any after adulthood Asthma patients who need bronchodilator for medical intervention can not be included).
8. Subjects with grade II or higher myocardial ischemia or myocardial infarction, and poorly controlled arrhythmias (including QTc interval ≥450ms in men and ≥470ms in women). According to the New York Heart Association standard, Subjects with grade III-IV cardiac insufficiency, or echocardiography showed left ventricular ejection fraction (LVEF) <50%; myocardial infarction occurred within 6 months before enrollment, and New York Heart Association grade II or above cardiac function Failure, uncontrolled angina, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, or electrocardiogram suggesting acute ischemia or active conduction system abnormalities.
9. Concurrent severe infection (eg, requiring intravenous antibiotics, antifungals, or antivirals) within 4 weeks prior to first dose, or unexplained fever >38.5°C during screening or before first dose.
10. Subjects with a history of psychotropic substance abuse and unable to quit or with mental disorders.
11. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA is higher than the detection limit of the analytical method) or co-infection with hepatitis B and C.
12. Subjects with untreated central nervous system metastases, Subjects who have received systemic, radical brain or meningeal metastases in the past (radiotherapy or surgery), have been stable for at least 1 month if confirmed by imaging, and have stopped systemic hormone therapy (Dose > 10mg/day prednisone or other equivalent therapeutic hormones) for more than 2 weeks and without clinical symptoms can be included.
13. Subjects with a history of hereditary or acquired bleeding or coagulation dysfunction (the investigator will determine whether they can be included).
14. Other conditions not considered suitable for inclusion by the researcher.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
3-year OS rate | 36 months
  Patient proportion to survival in the third year

SECONDARY OUTCOMES:
Progression-free survival（PFS） | 24 months
  The period of time between when a patient with neoplastic disease receives treatment and when the disease progresses or death from any cause occurs.
Objective response rate (ORR) | 12 months
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including cases of complete remission（CR） and partial remission（PR）.
Acute Adverse Events (AEs) | 36 months
  The number of participants who experience unacceptable toxicity during protocol treatment as measured by the NCI CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China